CLINICAL TRIAL: NCT02276417
Title: Persistent Inflammation, Immunosuppression and Catabolism Syndrome (PICS): A New Horizon for Surgical Critical Care Subtitle: Cardiac Dysfunction in Older Sepsis Survivors Subtitle: Development of a Designer Proline-Rich Antimicrobial Peptide Chaperone Protein Inhibitor (DPC) for Treating Sepsis
Brief Title: PICS: Subtitle Cardiac Dysfunction in Older Sepsis Survivors
Acronym: PICS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400611-N; P50GM111152-01 (NIH); OCR14760 (Other: Universiy of Florida)
Record Dates: First submitted 2014-10-15; First posted 2014-10-28 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2024-12

CONDITIONS: Sepsis
Keywords: Sepsis; Surgical ICU
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Blood Collection. Urine collection. Bioimpedance analysis. Quality-of-life questionnaires, physical function tests and cognitive function tests.
  Interventions: Other: Blood collection; Other: Urine collection; Other: Bioimpedance Analysis; Other: Cognitive Function Tests; Other: Quality-of-life Questionnaires; Other: Physical Function Tests
- Healthy Controls: Blood Collection.
  Interventions: Other: Blood Collection

INTERVENTIONS:
Other: Blood collection — Blood will be collected from patient at baseline, day 1, day 4, day 7 and weekly until week 6 as long as the patient is still hospitalized. Blood will also be collected at the one year appointment.
  Groups: Sepsis
Other: Urine collection — Urine will be collected from patient at baseline, day 1, day 4, day 7 and weekly until week 6 as long as the patient is still hospitalized. Urine will also be collected at the one year appointment.
  Groups: Sepsis
Other: Bioimpedance Analysis — The bioimpedance analysis will be performed at baseline, day 14 or discharge from hospitalization, month 3, month 6, and month 12.
  Other Names: BIA
  Groups: Sepsis
Other: Cognitive Function Tests — Cognitive function tests will be administered at 3, 6 and 12 months.
  Groups: Sepsis
Other: Quality-of-life Questionnaires — Quality-of-life questionnaires will be administered at baseline, 3, 6 and 12 months.
  Groups: Sepsis
Other: Physical Function Tests — Physical function tests will be administered at baseline, day 14 or discharge from hospital 3, 6 and 12 months.
  Groups: Sepsis
Other: Blood Collection — The healthy volunteer participants will donate a blood sample. These controls will allow the investigators to determine if the values obtained are accurate, reliable, and repeatable.
  Groups: Healthy Controls

SUMMARY:
The purpose of this study is to define the natural history and causes of chronic critical illness (CCI) in surgical intensive care patients who have had sepsis. The investigator also wants to define the long-term physical and cognitive outcomes of this disease. The investigator will be looking at many clinical variables to try to define CCI.

DETAILED DESCRIPTION:
This is a prospective, observational study aimed at identifying the frequency, natural history and long term outcomes of CCI and PICS in the survivors of surgical or trauma-associated sepsis.

A major portion of the translational data to be obtained will be from urine and blood samples from septic patients identified in the surgery and trauma ICUs. The blood will be processed for genomic markers, inflammatory markers, immunosuppression markers, Myeloid Derived Suppressor Cells (MDSC) functions, and angiogenic factors. The urine will be processed for messenger RNA (mRNA) isolation and protein biomarkers.

Bioimpedance analysis will performed to assess body composition. In order to assess the long term outcomes, the following Quality-of-life, functional and cognitive tests will be performed.

Health-related quality of life questionnaire, EuroQol-5D, Mini Nutritional Assessment Form, the Hopkins Verbal Learning Test, Controlled Oral Word Association, Modified Mini-Mental Status Exam, Short PhysicalPerformance Battery, Hand Grip Strength Measurement and The Eastern Cooperative Oncology Group (ECOG), World Health Organization (WHO), Zubrod Scale Healthy volunteer subjects will be identified from the general population. Healthy subjects will be screened via inclusion/exclusion criteria upon contact. If appropriate for participation, the subject will be consulted for consent.

ELIGIBILITY:
Inclusion Criteria:

* presence in the surgery or trauma intensive care unit (ICU) at University of Florida (UF) Health Shands Hospital where clinical care can be managed by surgical critical care guided by standard operating procedures.
* age of ≥18 years
* placed on EMR sepsis protocol with sepsis/septic shock by Sepsis-3 criteriad
* ability to obtain informed consent.

Exclusion Criteria:

* patients deemed to be futile care or have advanced care directives or goals of care limiting resuscitative efforts.
* severe traumatic brain injury (evidence of neurologic injury on CT scan and a Glasgow Coma Scale (GCS) <8 after resuscitation).
* refractory shock (i.e., patients who die within 12 hours).
* uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel)
* severe Congestive Heart Failure (CHF) (NY Heart Association Class IV)
* severe chronic liver disease (Childs-Pugh Class B/C and /or MELD > 14) or pre-liver transplant.
* known HIV infection with CD4 count <200 cells/mm3
* organ transplant recipient on immunosuppressive agents
* known pregnancy
* prisoners
* institutionalized patients
* inability to obtain informed consent.
* pre-hospital bedridden status (WHO/Zubrod score ≥ 4).
* patient's with an exacerbation of historic CVD or new onset CVD
* alternative or confounding diagnosis causing shock state (e.g. MI or PE)
* enrollment > 96 hours after suspected sepsis onset.
* pre-existing state of Chronic critical illness (ICU LOS ≥ 14 days, includes outside facility)
* interfacility transfer patients with > 96 hour critical illness prior to transfer.
* subsequent clinical adjudication not consistent with sepsis/septic shock by Sepsis-3 criteria

Healthy Controls

Inclusion criteria will be:

* all adults (age ≥18)
* Ability to obtain Informed Consent prior to blood collection.

Exclusion Criteria will be:

* Current, chronic steroid use
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are looking at all patients admitted to the surgical and trauma ICUs that have been entered into the sepsis protocol.
Sampling Method: Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
A change in the results in blood markers for persistent inflammatory state from baseline, Day 1, Day 4, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, and one year. | Baseline, Day 1, Day 4, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, and one year.
  Participant's blood will be analyzed for a persistent inflammatory state, anemia and adaptive immunosuppression. To look at whether sepsis alters the angiogenic balance between angiotensin II (ANGII), erythropoietin, and the VEGF receptor (VEGFR), and whether this imbalance is required for myeloid-derived suppressor cell (MDSC) expansion and chronic critical illness (CCI) and catabolism syndrome (PICS) development.
A change in the results for mRNA isolation and protein biomarkers from baseline, Day 1, Day 4, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, and one year. | Baseline, Day 1, Day 4, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, and one year.
  The urine will be processed for mRNA isolation and protein biomarkers.
A change in the results of the Dys-HDL baseline to day 4 | Baseline and Day 4
  Participant's blood will be analyzed to extensively characterize the temporal relationship between Dys-HDL, pertinent enzymes, and sepsis and endothelial biomarkers in patients with sepsis.

SECONDARY OUTCOMES:
A change in results from the Hopkins Verbal Learning Test from 3 months, 6 months and one year. | 3 months, 6 months and one year.
  A 12-item learning and memory test designed for brief, easy administration with proven participant tolerability in a variety of populations. The highest score is 36 and the lowest score is 12. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in results from the Controlled Oral Word Association from 3 months, 6 months and one year. | 3 months, 6 months and one year.
  Measures executive function and verbal fluency. Patients are asked to generate as many words as possible beginning with specific letters. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
a change iin the results from the Modified Mini-Mental Status Exam from 3 months, 6 months and one year. | 3 months, 6 months and one year.
  A measure of global cognitive functioning. This is an expanded 100- point version of the original Folstein Modified Mini-Mental Status Exam. A score greater than or equal to 27 overall points indicates a normal cognition, below this score can indicate severe (-9), moderate (10-18) or mild (19 -24) cognitive impairment. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results form the Health-related Quality of Life questionnaire from baseline, 3 months, 6 months and one year. | Baseline, 3 months, 6 months and one year.
  The Medical Outcome Study 36-item short form (SF-36) is a measure of health-related quality of life (HRQOL). It scores eight domains of health: physical functioning, role limitations due to physical health, role limitations due to emotional problems, vitality (energy/fatigue), mental health, bodily pain, social functioning, and general health perceptions on a scale from 0 to 100, with 100 representing the highest level of functioning possible. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results from the EuroQol-5D (EQ-5D) questionnaire from baseline, 3 months, 6 months and one year. | Baseline, 3 months, 6 months and one year.
  The EQ-5D is an HRQOL instrument with established validity in critical care survivors and as a surrogate-completed proxy measure. This tool is a descriptive system of health-related quality-of-life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of three responses. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results of the Mini Nutritional Assessment Form (MNA-SF) baseline, 3 months, 6 months and one year. | Baseline, 3 months, 6 months and one year.
  This is a validated nutrition screening and assessment tool that can identify patients who are malnourished or at risk for malnutrition. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results of the Short Physical Performance Battery from 3 months, 6 months and one year. | 3 months, 6 months and one year.
  Based on a timed short-distance (4 min) walk, repeated chair stands, and balance test. A score of 0 to 4 will be determined for each component, and a summary score ranging from 0 (worst performers) to 12 (best performers) will be calculated. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results of the Hand Grip Strength Measurement from baseline, day 14 or discharge from hospital, 3 months, 6 months and one year. | baseline, 14 days or hospital discharge, 3 months, 6 months and one year.
  Using an adjustable, hydraulic grip strength dynamometer. Three trials will be conducted for each hand. The best performance for each hand will be recorded. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results from The ECOG/WHO/Zubrod Scale from 3 months, 6 months and one year. | 3 months, 6 months and one year.
  A 5-point scale that measures the performance status of a patient's ambulatory nature: 0) Asymptomatic (fully active), 1) Symptomatic but completely ambulatory (restricted in physically strenuous activity), 2) Symptomatic, <50% in bed during the day (ambulatory and capable of all selfcare but unable to perform any work activities), 3) Symptomatic, >50% in bed, but not bedbound (capable of only limited self-care), 4) Bedbound (completely disabled, incapable of any self-care), and 5) Death. The test will be performed to look at the epidemiology and long-term physical and cognitive outcomes of chronic critical illness (CCI) in surgical intensive care unit (ICU) participants who survive sepsis.
A change in the results from the Bioimpedance analysis from baseline, day 14 or hospital discharge, 3 months, 6 months, and one year. | baseline, 14 days or hospital discharge, 3 months, 6 months, and one year.
  Using a Biodynamics BIA 450 to measure the content of water, muscle and fat to assess body composition

OTHER OUTCOMES:
Mortality | Up to one year
  Mortality will be assessed daily while the subject is in the hospital and then at post discharge follow up visits or by phone if the subject is unable to come to the follow up appointments. The Social Security mortality database will be accessed for subjects that are lost to follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Efron, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital, Gainesville, Florida, United States

REFERENCES:
- [Derived] Barrios EL, Balzano-Nogueira L, Polcz VE, Rodhouse C, Leary JR, Darden DB, Rincon JC, Dirain ML, Ungaro R, Nacionales DC, Larson SD, Sharma A, Upchurch G, Wallet SM, Brusko TM, Loftus TJ, Mohr AM, Maile R, Bacher R, Cai G, Kladde MP, Mathews CE, Moldawer LL, Brusko MA, Efron PA. Unique lymphocyte transcriptomic profiles in septic patients with chronic critical illness. Front Immunol. 2024 Dec 3;15:1478471. doi: 10.3389/fimmu.2024.1478471. eCollection 2024. PMID 39691721
- [Derived] Barrios EL, Rincon JC, Willis M, Polcz VE, Leary JR, Darden DB, Balch JA, Larson SD, Loftus TJ, Mohr AM, Wallet S, Brusko MA, Balzano-Nogueira L, Cai G, Sharma A, Upchurch GR Jr, Kladde MP, Mathews CE, Maile R, Moldawer LL, Bacher R, Efron PA. TRANSCRIPTOMIC DIFFERENCES IN PERIPHERAL MONOCYTE POPULATIONS IN SEPTIC PATIENTS BASED ON OUTCOME. Shock. 2024 Aug 1;62(2):208-216. doi: 10.1097/SHK.0000000000002379. Epub 2024 May 2. PMID 38713581
- [Derived] Stortz JA, Cox MC, Hawkins RB, Ghita GL, Brumback BA, Mohr AM, Moldawer LL, Efron PA, Brakenridge SC, Moore FA. Phenotypic heterogeneity by site of infection in surgical sepsis: a prospective longitudinal study. Crit Care. 2020 May 7;24(1):203. doi: 10.1186/s13054-020-02917-3. PMID 32381107
- [Derived] Hollen MK, Stortz JA, Darden D, Dirain ML, Nacionales DC, Hawkins RB, Cox MC, Lopez MC, Rincon JC, Ungaro R, Wang Z, Wu Q, Brumback B, Gauthier ML, Kladde M, Leeuwenburgh C, Segal M, Bihorac A, Brakenridge S, Moore FA, Baker HV, Mohr AM, Moldawer LL, Efron PA. Myeloid-derived suppressor cell function and epigenetic expression evolves over time after surgical sepsis. Crit Care. 2019 Nov 13;23(1):355. doi: 10.1186/s13054-019-2628-x. PMID 31722736
- [Derived] Brakenridge SC, Moore FA, Mercier NR, Cox M, Wu Q, Moldawer LL, Mohr AM, Efron PA, Smith RS. Persistently Elevated Glucagon-Like Peptide-1 Levels among Critically Ill Surgical Patients after Sepsis and Development of Chronic Critical Illness and Dismal Long-Term Outcomes. J Am Coll Surg. 2019 Jul;229(1):58-67.e1. doi: 10.1016/j.jamcollsurg.2019.04.014. Epub 2019 Apr 13. PMID 30991107
- [Derived] Gardner AK, Ghita GL, Wang Z, Ozrazgat-Baslanti T, Raymond SL, Mankowski RT, Brumback BA, Efron PA, Bihorac A, Moore FA, Anton SD, Brakenridge SC. The Development of Chronic Critical Illness Determines Physical Function, Quality of Life, and Long-Term Survival Among Early Survivors of Sepsis in Surgical ICUs. Crit Care Med. 2019 Apr;47(4):566-573. doi: 10.1097/CCM.0000000000003655. PMID 30664526
- [Derived] Stortz JA, Mira JC, Raymond SL, Loftus TJ, Ozrazgat-Baslanti T, Wang Z, Ghita GL, Leeuwenburgh C, Segal MS, Bihorac A, Brumback BA, Mohr AM, Efron PA, Moldawer LL, Moore FA, Brakenridge SC. Benchmarking clinical outcomes and the immunocatabolic phenotype of chronic critical illness after sepsis in surgical intensive care unit patients. J Trauma Acute Care Surg. 2018 Feb;84(2):342-349. doi: 10.1097/TA.0000000000001758. PMID 29251709